CLINICAL TRIAL: NCT02386787
Title: Ultrasound Assessment of Gastric Content for Semi Emergency Surgery
Acronym: ECHO-GAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1308170; 2013-A01649-36 (Other: ANSM)
Record Dates: First submitted 2015-02-20; First posted 2015-03-12 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-03

CONDITIONS: Anesthesia; Surgical Procedure, Unspecified
Keywords: Ultrasonography; Non-elective surgery; Anesthesia
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SEMI EMERGENCY SURGERY PATIENT (Experimental): patient undergoing a non-elective surgery and having a preoperative fasting period of six hours.
  Interventions: Device: Ultrasonography

INTERVENTIONS:
Device: Ultrasonography — an ultrasonography will be conducted before the anesthesic procedure to provide reliable quantitative information about the volume of gastric content.

SUMMARY:
Aspiration of gastric content is a rare but serious complication of anesthesia. In this context, preoperative fasting for elective surgery is well defined. In an emergency situation, international guidelines recommend rapid sequence of anesthesia to reduce the risk of aspiration. In semi emergency situation, there is no consensus about the anesthetic procedure even if a preoperative fasting has been observed due to uncertainty of gastric emptying related to stress or painful condition. The choice of anesthesia induction technique depends mainly on the anesthetist. Ultrasonography is a non invasive bedside tool that can provide reliable quantitative information about the volume of gastric content.

ELIGIBILITY:
Inclusion Criteria:

* undergoing a non-elective surgery
* having a preoperative fasting period of six hours

Exclusion Criteria:

* patients with digestive diseases (gastroesophageal reflux disease, hiatal hernia, active peptic ulcer, upper gastrointestinal bleeding, vagal denervation, pyloric stenosis, extrinsic digestive compression, occlusive syndrome), neurologic diseases (spinal cord injury over T10, amylose, Shy-Drager syndrome)
* patients with full stomach (preoperative fasting under 6 hours),
* pregnant women (over 15 weeks of amenorrhea)
* patients who received premedication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
patients with full stomach | baseline
  Full stomach is defined by an antral cross-section area (CSA) > 410 mm2, measured by ultrasonography

SECONDARY OUTCOMES:
duration of preoperative fasting | baseline
type of surgery disease | baseline
preoperative pain | baseline
  Visual Analog Scale
feeling of hunger | baseline
nausea and vomiting | baseline
  number of patients with nausea and vomiting
type of anesthetic procedure performed | baseline
  rapid or standard anesthetic induction
inhalation of gastric contents | baseline
  number of patients with inhalation of gastric contents during intervention

CONTACTS AND LOCATIONS:
Overall Officials: Julie GAVORY, MD, Principal Investigator — CHU de Saint Etienne
Locations (1):
- Chu de Saint Etienne, Saint-Etienne, France